CLINICAL TRIAL: NCT04151914
Title: Prevalence of Auditory Dysfunction and ICU-acquired Delirium Following Cardiac Surgery With Cardiopulmonary Bypass: a Prospective Observational Study
Acronym: AUDICS-ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Georges Pompidou Hospital (Other)
Responsible Party: Principal Investigator, Matthieu Daniel, Principal Investigator, European Georges Pompidou Hospital
Other Study IDs: AUDICS-ICU
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Hearing Loss; Cardiac Surgery; Cardiopulmonary Bypass; Postoperative Cognitive Dysfunction; Delirium
MeSH Terms: conditions — Hearing Loss; Postoperative Cognitive Complications; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
AUDICS-ICU is a prospective observational aiming to evaluate the prevalence of auditive dysfunction following cardiac surgery. Participants will undergo audiometric testings before and 3 months after cardiac surgery with cardiopulmonary bypass. Furthermore, the study evaluates hearing loss-associated ICU-acquired delirium after cardiac surgery with cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Undergoing non urgent cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Pregnant
* History of ear surgery
* Ear disease
* Inadequate understanding of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Over 18 years old undergoing non urgent cardiac surgery with cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of auditive dysfunction following cardiac surgery with cardiopulmonary bypass | 3 months
  Change from baseline audiometric testings at 3 months after cardiac surgery with cardiopulmonary bypass

SECONDARY OUTCOMES:
ICU-acquired delirium | 7 days
  Diagnose by CAM-ICU scale during ICU stay (if positive meaning the patient has delirium, CAM-ICU negative meaning the patient doesn't have delirium)
Cerebral perfusion | 7 days
  Near infrared spectroscopy during per operative period and transcranial doppler during ICU stay
Patient's quality of life after cardiac surgery: Survey | 3 months
  Survey evaluation quality of life at the end of ICU stay (IPREA) and 3 months after surgery. On a scale from 0 (best quality of life) to 100 (low quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Daniel, MD, Principal Investigator — European George Pompidou Hospital; Bernard Cholley, PHD, Study Director — European George Pompidou Hospital
Locations (1):
- Georges Pompidou European Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No